CLINICAL TRIAL: NCT05424380
Title: A Phase 1, Open Label Study of Intravenous GSK3745417 to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Determine RP2D and Schedule in Participants With Relapsed or Refractory Myeloid Malignancies Including Acute Myeloid Leukemia (AML) and High-risk Myelodysplastic Syndrome (HR-MDS)
Brief Title: A Phase 1, Open Label Study of Intravenous GSK3745417 to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Determine RP2D & Schedule in Participants With Relapsed or Refractory Myeloid Malignancies Including AML and HR MDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The protocol was terminated on the basis of a reprioritization of organizational allocation of resources for clinical research programs.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209809
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: GSK3745417; Acute myeloid leukemia; AML; high-risk myelodysplastic syndrome; HR-MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose escalation (Experimental): Part 1 will evaluate a dosing schedule for a total of 28 days in each cycle. The starting dose for Cycle 1 will be escalated in the next dose escalation cohort until MTD is reached.
  Interventions: Drug: GSK3745417
- Part 2: Dose expansion (Experimental): Part 2 will evaluate efficacy after an induction phase. The induction phase consists of a treatment regimen at RP2D determined in Part 1.
  Interventions: Drug: GSK3745417

INTERVENTIONS:
Drug: GSK3745417 — GSK3745417 will be administered

SUMMARY:
This is a Phase 1, open label, two-part study to determine recommended phase 2 dose (RP2D) and schedule of GSK3745417 administration in participants with relapsed/refractory AML or HR-MDS.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age and ≤75 years of age at the time of signing the informed consent for dose escalation and >18 years of age at the time of signing the informed consent for the dose expansion.
* Participants must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants with AML/HR MDS are eligible for participation in Part 1 and Part 2 if they have:

  1. A diagnosis of AML according to the World Health Organization 2016 criteria with relapsed or refractory disease and ineligible for or have exhausted standard therapeutic options.
  2. Have high-risk or high/very high by Revised International Prognostic Scoring System (IPSS-R) for MDS (restricted to Part 1) that has relapsed after or been refractory to prior therapy with hypomethylating agent.
* Participants with a prior history of stem cell transplant (autologous and/or allogeneic) are allowed if:

No clinical signs or symptoms of graft versus host disease (other than Grade 1 GVHD (<25% skin surface affected) and the participant is off all systemic immunosuppression. (Note: topical steroids for G1 skin GVHD are permitted on study)

* Participants must agree to abide by the gender specific contraceptive requirements below:

Female participants are eligible to participate if they are not either pregnant or breastfeeding, and at least one of the following conditions applies:

1. Is not a woman of childbearing potential (WOCBP), or
2. Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), The effectiveness of the contraceptive method will be evaluated by the investigator in relationship to the first dose of study treatment.

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APML or t(15;17) PML-RARA fusion). Patients with biphenotypic disease are excluded.
* Active central nervous system (CNS) involvement or disorder; and well controlled with ongoing treatment
* Participants with Immediate life-threatening, severe complications of leukemia (sepsis, hemorrhage).
* Participants with extramedullary disease as the sole site of AML
* Participants with active severe or uncontrolled infection,
* Participants with active autoimmune disease that has required systemic disease modifying or immunosuppressive treatment within the last 2 years.
* Participants with concurrent medical condition requiring the use of systemic immunosuppressive treatment within 28 days before the first dose of study treatment.
* Participants with history of vasculitis at any time prior to study treatment.
* Participant with a history of other malignancies less than 2 years prior to study entry,
* Participants with QT interval corrected using Fridericia's formula (QTcF) >450 millisecond (msec) for male participants, >470 msec for female participants, or >480 msec for participants with bundle branch block.
* Participants with recent history of allergen desensitization therapy within 4 weeks of starting study treatment.
* Participants with history or evidence of cardiovascular (CV) risk history of immune myocarditis or pericarditis.
* Participants with prior STING therapy.
* Participants with prior solid organ transplantation.
* Participants with recent prior therapy defined as follows: any non-monoclonal anti-cancer therapy within 14 days or 5 half-lives, whichever is longer, prior to start of study treatment; prior therapy with biological agents (including monoclonal antibodies) within 28 days prior to start of study treatment; any radiotherapy or major surgery within 14 days prior to start of study treatment; currently receiving investigational therapy in a clinical trial
* Participants with immune-related toxicity related to prior treatment that has not resolved to Grade ≤1 (except alopecia, hearing loss or Grade ≤2 neuropathy or endocrinopathy managed with replacement therapy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- GSK Investigational Site, Toronto, Ontario, Canada
- Germany (2):
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Leipzig
- Italy (3):
  - GSK Investigational Site, Meldola FC
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Roma
- GSK Investigational Site, Rotterdam, Netherlands
- Spain (2):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study conducted in a staged approach consisting of 2 parts. This study was terminated due to termination of asset after Part 1. Hence, no participants were enrolled in Part 2 of the study.
Pre-assignment Details: A total of 18 participants were enrolled in Part 1 of the study.
Groups:
- Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug: Participants with relapsed or refractory acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (HR-MDS) received GSK3745417 12.5 microgram (ug), powder for solution as intravenous (IV) injection from Days 1 to 28 (Cycle 1) followed by GSK3745417 25 ug, powder for solution as IV injection from Days 29 to 57 (Cycle 2); further followed by GSK3745417 50 ug, powder for solution as IV injection from Days 58 to 86 (Cycle 3). Each cycle was of 28 days.
- Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug: Participants with relapsed or refractory AML and HR-MDS received GSK3745417 25 ug, powder for solution as IV injection from Days 1 to 28 (Cycle 1) followed by GSK3745417 50 ug, powder for solution as IV injection from Days 29 to 57 (Cycle 2); further followed by GSK3745417 100 ug, powder for solution as IV injection from Days 58 to 86 (Cycle 3). Each cycle was of 28 days.
- Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug: Participants with relapsed or refractory AML and HR-MDS received GSK3745417 50 ug, powder for solution as IV injection from Days 1 to 28 (Cycle 1) followed by GSK3745417 100 ug, powder for solution as IV injection from Days 29 to 57 (Cycle 2); further followed by GSK3745417 200 ug, powder for solution as IV injection from Days 58 to 86 (Cycle 3). Each cycle was of 28 days.
- Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug: Participants with relapsed or refractory AML and HR-MDS received GSK3745417 100 ug, powder for solution as IV injection from Days 1 to 28 (Cycle 1) followed by GSK3745417 200 ug, powder for solution as IV injection from Days 29 to 57 (Cycle 2); further followed by GSK3745417 300 ug, powder for solution as IV injection from Days 58 to 86 (Cycle 3). Each cycle was of 28 days.
- Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug: Participants with relapsed or refractory AML and HR-MDS received GSK3745417 200 ug, powder for solution as IV injection from Days 1 to 28 (Cycle 1) followed by GSK3745417 300 ug, powder for solution as IV injection from Days 29 to 57 (Cycle 2); further followed by GSK3745417 300 ug, powder for solution as IV injection from Days 58 to 86 (Cycle 3). Each cycle was of 28 days.
- Part 2: GSK3745417: Participants in Part 2 with relapsed or refractory AML and HR-MDS were planned to receive GSK3745417 starting at the maximum tolerated dose determined from Part 1 of the study.
Period: Part 1: Cohort 1: 12.5 ug (Days 1 to 28)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 4 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Cohort 1: 25 ug (Days 29 to 57)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 3 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Cohort 1: 50 ug (Days 58 to 86)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 2 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Cohort 2: 25 ug (Days 1 to 28)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 1: Cohort 2: 50 ug (Days 29 to 57)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Cohort 2: 100 ug (Days 58 to 86)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 1: Cohort 3: 50 ug (Days 1 to 28)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Cohort 3: 100 ug (Days 29 to 57)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 1: Cohort 3: 200 ug (Days 58 to 86)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 1 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 1: Cohort 4:100 ug (Days 1 to 28)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 1: Cohort 4: 200 ug (Days 29 to 57)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 0 | 2 | 0 | 0
Completed | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 1: Cohort 4: 300 ug (Days 58 to 86)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 0 | 1 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 1: Cohort 5: 200 ug (Days 1 to 28)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 0 | 0 | 5 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 1: Cohort 5: 300 ug (Days 29 to 57)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 0 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Cohort 5: 300 ug (Days 58 to 86)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 0 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 2 (Up to 49 Weeks)
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417
Started | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated due to termination of asset after Part 1. Hence, no participants were enrolled in Part 2 of the study and data was not collected for Part 2 of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 1: GSK3745417 12.5 ug Followed by 25 ug Followed by 50 ug | Part 1: Cohort 2: GSK3745417 25 ug Followed by 50 ug Followed by 100 ug | Part 1: Cohort 3: GSK3745417 50 ug Followed by 100 ug Followed by 200 ug | Part 1: Cohort 4: GSK3745417 100 ug Followed by 200 ug Followed by 300 ug | Part 1: Cohort 5: GSK3745417 200 ug Followed by 300 ug Followed by 300 ug | Part 2: GSK3745417 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 5 | 0 | 18
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 44.0 (17.11) | 71.3 (4.73) | 69.7 (4.04) | 53.7 (15.31) | 67.0 (7.07) |  | 60.8 (14.69)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 2 |  | 8
  Male | 2 | 1 | 2 | 2 | 3 |  | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 |  | 0
  Not Hispanic or Latino | 4 | 3 | 3 | 3 | 5 |  | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-emergent (TE) Adverse Events (AEs) and TE Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involved medical or scientific judgment. A TEAE is an event that emerges during treatment having been absent pretreatment or worsens relative to the pretreatment state.
Time Frame: Up to 11.3 weeks
Population: Safety Population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: GSK3745417 12.5 ug: Participants with relapsed or refractory AML and HR-MDS received 12.5 ug GSK3745417 powder for solution as IV injection.
- Part 1: GSK3745417 25 ug: Participants with relapsed or refractory AML and HR-MDS received 25 ug GSK3745417 powder for solution as IV injection.
- Part 1: GSK3745417 50 ug: Participants with relapsed or refractory AML and HR-MDS received 50 ug GSK3745417 powder for solution as IV injection.
- Part 1: GSK3745417 100 ug: Participants with relapsed or refractory AML and HR-MDS received 100 ug GSK3745417 powder for solution as IV injection.
- Part 1: GSK3745417 200 ug: Participants with relapsed or refractory AML and HR-MDS received 200 ug GSK3745417 powder for solution as IV injection.
- Part 1: GSK3745417 300 ug: Participants with relapsed or refractory AML and HR-MDS received 300 ug GSK3745417 powder for solution as IV injection.
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 100 ug | Part 1: GSK3745417 200 ug | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 4 | 6 | 6 | 8 | 8 | 2
Participants
  TEAEs | 4 | 6 | 5 | 8 | 8 | 2
  TESAEs | 4 | 4 | 1 | 5 | 5 | 1

2. Primary Outcome: Part 1: Number of Participants With TEAEs and TESAEs by Severity Grades
Description: AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involved medical or scientific judgment. TEAE is an event that emerges during treatment having been absent pretreatment or worsens relative to the pretreatment state. AEs were graded by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) (version 5.0): Grade(G) 1=Mild, G2=Moderate, G3=Severe or medically significant but not immediately life-threatening, G4=Life-threatening consequences, G5=Death related AE.
Time Frame: Up to 11.3 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 100 ug | Part 1: GSK3745417 200 ug | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 4 | 6 | 6 | 8 | 8 | 2
Participants
  TEAEs, Grade 1 | 0 | 0 | 0 | 1 | 1 | 0
  TEAEs, Grade 2 | 0 | 2 | 2 | 0 | 1 | 0
  TEAEs, Grade 3 | 3 | 1 | 1 | 6 | 3 | 1
  TEAEs, Grade 4 | 1 | 1 | 2 | 0 | 2 | 1
  TEAEs, Grade 5 | 0 | 2 | 0 | 1 | 1 | 0
  TESAEs, Grade 1 | 0 | 1 | 1 | 1 | 0 | 0
  TESAEs, Grade 2 | 1 | 0 | 0 | 0 | 1 | 0
  TESAEs, Grade 3 | 3 | 1 | 0 | 3 | 2 | 1
  TESAEs, Grade 4 | 0 | 0 | 0 | 0 | 1 | 0
  TESAEs, Grade 5 | 0 | 2 | 0 | 1 | 1 | 0

3. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLT)
Description: An AE is considered to be a DLT if it is considered by the investigator to be clinically relevant and attributed (definitely, probably, or possibly) to the study intervention and meets at least 1 of the criteria listed below. Criteria for DLT included Grade(G)3 or 4 Cytokine Release Syndrome (CRS); G3 or 4 tumor lysis syndrome (TLS) that cannot be managed/ is not resolved within 72 hours (h); Liver Toxicity included Alanine aminotransferase (ALT)>=3* upper limit of normal (ULN), plus bilirubin>=2* ULN (>35 percent [%] direct) or plus international normalized ratio (INR)>1.5 (Possible Hy's law); G>=3 non-hematologic toxicity of any duration; G>=3 immune-related toxicity that does not resolve to G<=1 or Baseline within 8 days despite adequate immune suppressive therapy. Any other event which in the judgment of the investigator and GSK Medical Monitor is considered to be a DLT.
Time Frame: Up to 28 days
Population: DLT-evaluable Population included all participants who took at least 1 dose of study intervention and followed for the DLT observation period or were withdrawn within the DLT observation period due to meeting the DLT criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 100 ug | Part 1: GSK3745417 200 ug | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 4 | 6 | 6 | 8 | 8 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 1: Number of Participants With Withdrawals Due to AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 11.3 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 100 ug | Part 1: GSK3745417 200 ug | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 4 | 6 | 6 | 8 | 8 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part 2: Objective Response Rate (ORR)
Description: Overall response rate (ORR) defined as the percentage of participants with a complete remission (CR), CR with incomplete platelet recovery (CRp), incomplete count recovery (CRi), or a partial remission (PR) as per response criteria for AML and HR-MDS. CR=The participant must achieve a morphologic leukemia-free state (<= 5% blasts) and have no evidence of extramedullary disease. The participant must be free of all symptoms related to leukemia, have an absolute neutrophil count >= 1*10^9/Liter (L) and platelet count >=100*10^9/L, and be transfusion independent. CRp: Marrow response as per CR but platelet count <100 × 10^9/L. CRi: Marrow response as per CR but platelet count <100*10^9/L or neutrophil count <1*10^9/L. PR=A decrease from Baseline of at least 50% in the number of bone marrow blasts, to between 5% and 25% of the bone marrow aspirate.
Time Frame: Up to Day 84
Population: Safety Population. No participants were enrolled in Part 2 of the study. Hence, data was not collected for Part 2 of the study.
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

6. Primary Outcome: Part 2: Number of Participants With TEAEs and TESAEs
Description: as for outcome 1
Time Frame: Up to 49 weeks
Population: as for outcome 5
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

7. Primary Outcome: Part 2: Number of Participants With TEAEs and TESAEs by Severity Grades
Description: AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involved medical or scientific judgment. TEAE is an event that emerges during treatment having been absent pretreatment or worsens relative to the pretreatment state. AEs were graded by the investigator according to NCI-CTCAE (version 5.0): G1=Mild, G2=Moderate, G3=Severe or medically significant but not immediately life-threatening, G4=Life-threatening consequences, G5=Death related AE.
Time Frame: Up to 49 weeks
Population: as for outcome 5
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

8. Primary Outcome: Part 2: Number of Participants With Dose Limiting Toxicities (DLT)
Description: An AE is considered to be a DLT if it is considered by the investigator to be clinically relevant and attributed (definitely, probably, or possibly) to the study intervention and meets at least 1 of the criteria listed below. Criteria for DLT included Grade(G)3 or 4 Cytokine Release Syndrome (CRS); G3 or 4 TLS that cannot be managed/ is not resolved within 72 hours (h); Liver Toxicity included ALT>=3*upper limit of normal (ULN), plus bilirubin>=2*ULN (>35% direct) or plus international normalized ratio (INR)>1.5 (Possible Hy's law); G>=3 non-hematologic toxicity of any duration; G>=3 immune-related toxicity that does not resolve to G<=1 or Baseline within 8 days despite adequate immune suppressive therapy. Any other event which in the judgment of the investigator and GSK Medical Monitor is considered to be a DLT.
Time Frame: Up to 28 days
Population: as for outcome 5
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

9. Primary Outcome: Part 2: Number of Participants With Withdrawals Due to AEs
Description: as for outcome 4
Time Frame: Up to 49 weeks
Population: as for outcome 5
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

10. Secondary Outcome: Part 1: Maximum Concentration (Cmax) Following Administration of GSK3745417 12.5 µg, 25 ug, 50 µg and 200 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30 and 45 minutes, 1, 2, 4, 6, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 4, 8, 24 hours on Day 5
Population: Pharmacokinetic (PK) Population included all participants from the Safety Analysis Set for whom a PK sample was obtained and analyzed. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 200 ug
Number analyzed (Participants) | 4 | 5 | 6 | 8
Nanogram/milliliter (ng/mL)
  DAY 1 | 4.0437 (63.1268) | 5.3407 (18.6391) | 11.4244 (15.6862) | 49.8671 (25.7641)
  DAY 5: number analyzed (Participants) | 3 | 5 | 4 | 5
  DAY 5 | 3.3922 (76.7856) | 9.9633 (50.2486) | 11.7986 (12.9766) | 55.8182 (32.3703)

11. Secondary Outcome: Part 1: Maximum Concentration (Cmax) Following Administration of GSK3745417 100 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30 and 45 minutes, 1, 2, 4, 6, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 1, 4, 8, 12, 24 hours on Day 5; Pre-dose, 5 minutes, 4, 8, 12 and 24 hours on Day 8; Pre-dose, 5 minutes, 4, 8 and 24 hours on Day 12
Population: Pharmacokinetic (PK) Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Part 1: GSK3745417 100 ug
Number analyzed (Participants) | 8
Nanogram/milliliter (ng/mL)
  DAY 1 | 23.4043 (34.9860)
  DAY 5: number analyzed (Participants) | 6
  DAY 5 | 27.9947 (33.7584)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 20.7000 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.
  DAY 12: number analyzed (Participants) | 2
  DAY 12 | 37.9700 (50.5418)

12. Secondary Outcome: Part 1: Maximum Concentration (Cmax) Following Administration of GSK3745417 300 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5 minutes, 1, 4, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 1, 4, 8, 12, 24 hours on Day 5; Pre-dose, 5 minutes, 4, 8, 24 hours on Day 8
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 2
Nanogram/milliliter (ng/mL)
  DAY 1 | 60.0576 (18.6563)
  DAY 5 | 83.6227 (13.7291)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 95.6000 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.

13. Secondary Outcome: Part 1: Area Under the Concentration-time Curve AUC(0-t) Following Administration of GSK3745417 12.5 µg, 25 µg, 50 µg and 200 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30 and 45 minutes, 1, 2, 4, 6, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 4, 8, 24 hours on Day 5
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 200 ug
Number analyzed (Participants) | 4 | 5 | 6 | 8
Hour*nanogram/milliliter (h*ng/mL)
  DAY 1 | 21.7427 (57.6324) | 18.3426 (105.4447) | 39.7661 (86.7711) | 115.7833 (86.2087)
  DAY 5: number analyzed (Participants) | 3 | 5 | 4 | 5
  DAY 5 | 24.5192 (70.8547) | 53.4229 (75.0209) | 40.3425 (46.5663) | 269.2527 (97.8566)

14. Secondary Outcome: Part 1: Area Under the Concentration-time Curve AUC(0-t) Following Administration of GSK3745417 100 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: GSK3745417 100 ug
Number analyzed (Participants) | 8
Hour*nanogram/milliliter (h*ng/mL)
  DAY 1 | 73.7605 (102.0968)
  DAY 5: number analyzed (Participants) | 6
  DAY 5 | 129.1817 (133.3992)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 88.3060 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.
  DAY 12: number analyzed (Participants) | 2
  DAY 12 | 246.3285 (273.1186)

15. Secondary Outcome: Part 1: Area Under the Concentration-time Curve AUC(0-t) Following Administration of GSK3745417 300 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 12
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 2
Hour*nanogram/milliliter (h*ng/mL)
  DAY 1 | 111.0980 (17.4746)
  DAY 5 | 156.7682 (21.7702)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 177.0957 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.

16. Secondary Outcome: Part 1: AUC (0-tau) Following Administration of GSK3745417 12.5 µg, 25 µg, 50 µg and 200 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30 and 45 minutes, 1, 2, 4, 6, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 4, 8, 24 hours on Day 5
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 200 ug
Number analyzed (Participants) | 4 | 5 | 6 | 8
Hour*nanogram/milliliter (h*ng/mL)
  DAY 1 | 22.0086 (58.5871) | 18.6671 (101.4660) | 40.4989 (86.3765) | 116.0595 (86.0517)
  DAY 5: number analyzed (Participants) | 3 | 5 | 4 | 5
  DAY 5 | 24.4250 (71.8245) | 53.6275 (75.3947) | 40.5395 (46.3785) | 267.9373 (98.1167)

17. Secondary Outcome: Part 1: AUC (0-tau) Following Administration of GSK3745417 100 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: GSK3745417 100 ug
Number analyzed (Participants) | 8
Hour*nanogram/milliliter (h*ng/mL)
  DAY 1 | 75.4673 (103.4499)
  DAY 5: number analyzed (Participants) | 6
  DAY 5 | 129.6654 (134.9177)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 88.4344 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.
  DAY 12: number analyzed (Participants) | 2
  DAY 12 | 247.2046 (272.2710)

18. Secondary Outcome: Part 1: AUC (0-tau) Following Administration of GSK3745417 300 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 12
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 2
Hour*nanogram/milliliter (h*ng/mL)
  DAY 1 | 111.2544 (17.7235)
  DAY 5 | 157.0654 (21.6207)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 177.2807 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.

19. Secondary Outcome: Part 1: AUC(0-infinity) Following Administration of GSK3745417 12.5 µg, 25 µg, 50 µg and 200 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30 and 45 minutes, 1, 2, 4, 6, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 4, 8, 24 hours on Day 5
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 200 ug
Number analyzed (Participants) | 4 | 5 | 6 | 8
Hour*nanogram/milliliter (h*ng/mL)
  DAY 1 | 24.1814 (58.7275) | 19.7396 (111.3832) | 44.1762 (110.0662) | 124.8946 (103.5148)
  DAY 5: number analyzed (Participants) | 3 | 5 | 4 | 5
  DAY 5 | 32.1932 (85.8221) | 61.4040 (89.9314) | 42.2109 (48.0113) | 302.1566 (119.5787)

20. Secondary Outcome: Part 1: AUC(0-infinity) Following Administration of GSK3745417 100 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: GSK3745417 100 ug
Number analyzed (Participants) | 8
Hour*nanogram/milliliter (h*ng/mL)
  DAY 1 | 82.4501 (122.0638)
  DAY 5: number analyzed (Participants) | 6
  DAY 5 | 149.6791 (171.2285)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 91.6906 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.
  DAY 12: number analyzed (Participants) | 1
  DAY 12 | 92.8915 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.

21. Secondary Outcome: Part 1: AUC(0-infinity) Following Administration of GSK3745417 300 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 12
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 2
Hour*nanogram/milliliter (h*ng/mL)
  DAY 1 | 113.4262 (17.3464)
  DAY 5 | 161.3749 (23.9753)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 179.2585 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.

22. Secondary Outcome: Part 1: Terminal Phase Elimination Rate Constant (Lambda Z) Following Administration of GSK3745417 12.5 µg, 25 µg, 50 µg and 200 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30 and 45 minutes, 1, 2, 4, 6, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 4, 8, 24 hours on Day 5
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 200 ug
Number analyzed (Participants) | 4 | 5 | 6 | 8
1/hour
  DAY 1 | 0.0958 (14.0287) | 0.1879 (122.9400) | 0.1614 (100.3767) | 0.1106 (98.3724)
  DAY 5: number analyzed (Participants) | 3 | 5 | 4 | 5
  DAY 5 | 0.0564 (23.4595) | 0.0902 (41.2921) | 0.1233 (7.5634) | 0.0924 (36.4027)

23. Secondary Outcome: Part 1: Terminal Phase Elimination Rate Constant (Lambda Z) Following Administration of GSK3745417 100 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Part 1: GSK3745417 100 ug
Number analyzed (Participants) | 8
1/hour
  DAY 1 | 0.1400 (114.8419)
  DAY 5: number analyzed (Participants) | 6
  DAY 5 | 0.0862 (43.9385)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 0.1300 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.
  DAY 12: number analyzed (Participants) | 2
  DAY 12 | 0.0603 (100.8393)

24. Secondary Outcome: Part 1: Terminal Phase Elimination Rate Constant (Lambda Z) Following Administration of GSK3745417 300 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 12
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 2
1/hour
  DAY 1 | 0.0978 (39.1392)
  DAY 5 | 0.1237 (39.1510)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 0.1512 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.

25. Secondary Outcome: Part 1: Terminal Phase Half-life (t1/2) Following Administration of GSK3745417 12.5 µg, 25 µg, 50 µg and 200 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30 and 45 minutes, 1, 2, 4, 6, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 4, 8, 24 hours on Day 5
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 200 ug
Number analyzed (Participants) | 4 | 5 | 6 | 8
Hour (h)
  DAY 1 | 7.2332 (14.0287) | 3.6895 (122.9400) | 4.2938 (100.3767) | 6.2658 (98.3724)
  DAY 5: number analyzed (Participants) | 3 | 5 | 4 | 5
  DAY 5 | 12.2931 (23.4595) | 7.6835 (41.2921) | 5.6202 (7.5634) | 7.4977 (36.4027)

26. Secondary Outcome: Part 1: Terminal Phase Half-life (t1/2) Following Administration of GSK3745417 100 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | Part 1: GSK3745417 100 ug
Number analyzed (Participants) | 8
Hour (h)
  DAY 1 | 4.9494 (114.8419)
  DAY 5: number analyzed (Participants) | 6
  DAY 5 | 8.0420 (43.9385)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 5.3318 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.
  DAY 12: number analyzed (Participants) | 2
  DAY 12 | 11.4948 (100.8393)

27. Secondary Outcome: Part 1: Terminal Phase Half-life (t1/2) Following Administration of GSK3745417 300 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 12
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 2
Hour (h)
  DAY 1 | 7.0877 (39.1392)
  DAY 5 | 5.6013 (39.1510)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 4.5845 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.

28. Secondary Outcome: Part 1: Systemic Clearance of Parent Drug (CL) Following Administration of GSK3745417 12.5 µg, 25 µg, 50 µg and 200 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30 and 45 minutes, 1, 2, 4, 6, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 4, 8, 24 hours on Day 5
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 200 ug
Number analyzed (Participants) | 4 | 5 | 6 | 8
Liter/hour (L/h)
  DAY 1 | 0.5169 (58.7275) | 1.2669 (110.9895) | 1.1313 (109.9904) | 1.5982 (103.1281)
  DAY 5: number analyzed (Participants) | 3 | 5 | 4 | 6
  DAY 5 | 0.3883 (85.8221) | 0.4090 (89.8847) | 1.1870 (48.4302) | 0.8532 (140.7702)

29. Secondary Outcome: Part 1: Systemic Clearance of Parent Drug (CL) Following Administration of GSK3745417 100 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | Part 1: GSK3745417 100 ug
Number analyzed (Participants) | 8
Liter/hour (L/h)
  DAY 1 | 1.2121 (121.9357)
  DAY 5: number analyzed (Participants) | 6
  DAY 5 | 0.6681 (171.2285)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 1.0906 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.
  DAY 12: number analyzed (Participants) | 2
  DAY 12 | 0.2935 (532.2277)

30. Secondary Outcome: Part 1: Systemic Clearance of Parent Drug (CL) Following Administration of GSK3745417 300 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 12
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 2
Liter/hour (L/h)
  DAY 1 | 2.6516 (17.5162)
  DAY 5 | 1.8769 (22.2726)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 1.6736 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.

31. Secondary Outcome: Part 1: Volume of Distribution (V) Following Administration of GSK3745417 12.5 µg, 25 µg, 50 µg and 200 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30 and 45 minutes, 1, 2, 4, 6, 8, 12, 24 hours on Day 1; Pre-dose, 5 minutes, 4, 8, 24 hours on Day 5
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 200 ug
Number analyzed (Participants) | 4 | 5 | 6 | 8
Liter (L)
  DAY 1 | 5.1242 (62.5343) | 6.1162 (15.1427) | 6.2318 (23.2325) | 7.2915 (35.8656)
  DAY 5: number analyzed (Participants) | 3 | 5 | 4 | 5
  DAY 5 | 7.9543 (44.7917) | 4.0818 (48.7367) | 6.7901 (18.9568) | 6.0176 (30.5236)

32. Secondary Outcome: Part 1: Volume of Distribution (V) Following Administration of GSK3745417 100 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Part 1: GSK3745417 100 ug
Number analyzed (Participants) | 8
Liter (L)
  DAY 1 | 6.8614 (41.4133)
  DAY 5: number analyzed (Participants) | 6
  DAY 5 | 6.2891 (42.2982)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 7.0024 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.
  DAY 12: number analyzed (Participants) | 2
  DAY 12 | 5.4797 (38.0866)

33. Secondary Outcome: Part 1: Volume of Distribution (V) Following Administration of GSK3745417 300 µg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 12
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Part 1: GSK3745417 300 ug
Number analyzed (Participants) | 2
Liter (L)
  DAY 1 | 7.9354 (16.5438)
  DAY 5 | 6.6325 (29.8240)
  DAY 8: number analyzed (Participants) | 1
  DAY 8 | 4.5465 (NA) — NA indicates data was not available as geometric coefficient of variation could not be calculated for a single participant.

34. Secondary Outcome: Part 2: Number of Participants With AEs, SAEs and Adverse Events of Special Interest (AESIs) Leading to Dose Modification and Dose Delays
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involved medical or scientific judgment. AESI includes events that were immune-related or related to Cytokine Release Syndrome or tumor lysis syndrome.
Time Frame: Up to 49 weeks
Population: as for outcome 5
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

35. Secondary Outcome: Part 2: Cmax Following Administration of GSK3745417
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: Pre-dose, 5, 15, 30, 45 minutes, 1, 2, 4, 6, 8, 12 and 24 hours on Day 1; Predose on Day 4; Pre-dose and 5 minutes, 4, 8, 24 hours on Day 5; Predose and 4, 8, 12 and 24 hours on Day 8; Pre-dose, 1, 4, 8, 12 and 24 hours on Day 12
Population: Pharmacokinetic (PK) Population. No participants were enrolled in Part 2 of the study. Hence, data was not collected for Part 2 of the study.
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

36. Secondary Outcome: Part 2: AUC(0-t) Following Administration of GSK3745417
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 35
Population: as for outcome 35
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

37. Secondary Outcome: Part 2: AUC(0-tau) Following Administration of GSK3745417
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 35
Population: as for outcome 35
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

38. Secondary Outcome: Part 2: AUC(0-infinity) Following Administration of GSK3745417
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 35
Population: as for outcome 35
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

39. Secondary Outcome: Part 2: Terminal Phase Elimination Rate Constant (Lambda Z) Following Administration of GSK3745417
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 35
Population: as for outcome 35
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

40. Secondary Outcome: Part 2: Terminal Phase Half-life (t1/2) Following Administration of Single Dose GSK3745417
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 35
Population: as for outcome 35
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

41. Secondary Outcome: Part 2: Systemic Clearance of Parent Drug (CL) Following Administration of GSK3745417
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 35
Population: as for outcome 35
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

42. Secondary Outcome: Part 2: Volume of Distribution (V) Following Administration of GSK3745417
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3745417.
Time Frame: as for outcome 35
Population: as for outcome 35
Arm/Group | Part 2: GSK3745417
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, treatment emergent (TE) non-serious adverse events (Non-SAEs) and TE serious adverse events (TESAEs) were collected up to 11.3 weeks in Part 1 of the study.
Description: Safety Population included all participants who take at least 1 dose of study intervention. This study was terminated due to termination of asset after Part 1. Hence, no participants were enrolled in Part 2 of the study and data was not collected for Part 2 of the study.
Arm/Group | Part 1: GSK3745417 12.5 ug | Part 1: GSK3745417 25 ug | Part 1: GSK3745417 50 ug | Part 1: GSK3745417 100 ug | Part 1: GSK3745417 200 ug | Part 1: GSK3745417 300 ug | Part 2: GSK3745417
All-Cause Mortality (participants affected / at risk) | 1/4 | 2/6 | 1/6 | 2/8 | 5/8 | 1/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/4 | 4/6 | 1/6 | 5/8 | 5/8 | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 3/4 | 5/6 | 5/6 | 7/8 | 8/8 | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK3745417 12.5 ug (N=4) | Part 1: GSK3745417 25 ug (N=6) | Part 1: GSK3745417 50 ug (N=6) | Part 1: GSK3745417 100 ug (N=8) | Part 1: GSK3745417 200 ug (N=8) | Part 1: GSK3745417 300 ug (N=2) | Part 2: GSK3745417 (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK3745417 12.5 ug (N=4) | Part 1: GSK3745417 25 ug (N=6) | Part 1: GSK3745417 50 ug (N=6) | Part 1: GSK3745417 100 ug (N=8) | Part 1: GSK3745417 200 ug (N=8) | Part 1: GSK3745417 300 ug (N=2) | Part 2: GSK3745417 (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT05424380/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT05424380/SAP_001.pdf